CLINICAL TRIAL: NCT03614871
Title: Snuff Use, Smoking, Periodontal Health and Premature Death: 30-year Study
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anna Julkunen, Principal Investigator, University of Helsinki
Other Study IDs: 00290
Record Dates: First submitted 2018-07-23; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Tobacco Use; Periodontitis
Keywords: Tobacco; Calculus; Gingiva; Oral hygiene; Periodontitis; Biofilm
MeSH Terms: conditions — Tobacco Use; Periodontitis; Calculi | interventions — Epidemiologic Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No arms: There are no interventions
  Interventions: Other: Epidemiological study

INTERVENTIONS:
Other: Epidemiological study

SUMMARY:
Snuff use and smoking associated with poor periodontal health, especially if used together.

DETAILED DESCRIPTION:
Aim: The investigators investigated how snuff use and smoking affect periodontal health parameters and mortality in a Swedish cohort, hypothesizing that snuff use increases the risks.

Material and methods: Study cohort of 1 532 subjects aged 30 to 40 (758 men and 774 women) from Stockholm area was clinically examined and followed up from 1985 to 2015. Associations were analysed between periodontal health parameters, snuff use, smoking and age of death. For analyses, all subjects were classified into four groups: "dual-users" (current and ex-snuffers, current and ex-smokers); "pure snuffers" (current and ex-snuffers); "pure smokers" (non-snuffers, current and ex-smokers) and "non-users" (non-snuffers and non-smokers). Cross-tabulation, chi-square and Fisher's exact tests were used.

ELIGIBILITY:
Inclusion Criteria:

* In 1985-1986 a sample was selected from the registry file of all inhabitants of the Stockholm area, of people born on the 20th of any month from 1945 to 1954.The sample comprised 3200 people. They were informed about the purpose of the study and called for clinical investigation. 1681 (52.5%) individuals, 840 men and 841 women, participated in the study. From the remaining 1519 non-respondents to the initial call, 100 randomly selected subjects, 45 men and 55 women, were reinformed and persuaded and finally agreed to participate in this investigation. They were used as a drop-out control sample.

Exclusion Criteria:

* Other people

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Swedish national database sample
Sampling Method: Probability Sample
Enrollment: 1676 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Periodontal Pockets | 1985
  Dual users, pure snuffers and pure smokers had more ≥5mm deep periodontal pockets than non-users. Periodontal pockets were measured from all teeth and from six surfaces with a Hu-Friedy (PCPUNC 15) periodontal probe (Hu-friedy, Chicago, Ill., USA).
Missing teeth | 1985
  Pure smokers had more likely missing teeth than subjects in other groups. Missing teeth were calculated my dentist in clinical examination.
Gingival Index (GI) | 1985
  Dual-users, pure snuffers and pure smokers had higher GI scores than non-users. GI was scored from 0 (no gum bleeding) to 3 (abundant gum bleeding)
Premature death | From year 1985 to year 2015
  Snuff users or smokers did not die earlier than non-users of the cohort in 30 years. The Swedish National Death Register listing the cumulated causes of all deaths was used in the analyses.
Plaque Index (PI) | 1985
  Dual-users, pure snuffers and pure smokers had higher PI scores than non-users. PI was scored from 0 (no plaque) to 3 (abundant plaque)
Calculus Index (CI) | 1985
  Dual-users, pure snuffers and pure smokers had higher CI scores than non-users. CI was scored from 0 (no calculus) to 3 (abundant calculus) according to Greene & Vermillion

IPD SHARING:
Plan to Share IPD: No
Any underlying research materials related to present study could be accessed by e-mail birgitta.soder@ki.se.

REFERENCES:
- [Background] Pihlstrom BL, Michalowicz BS, Johnson NW. Periodontal diseases. Lancet. 2005 Nov 19;366(9499):1809-20. doi: 10.1016/S0140-6736(05)67728-8. PMID 16298220
- [Background] Nibali L, Farias BC, Vajgel A, Tu YK, Donos N. Tooth loss in aggressive periodontitis: a systematic review. J Dent Res. 2013 Oct;92(10):868-75. doi: 10.1177/0022034513501878. Epub 2013 Aug 16. PMID 23955159
- [Background] Page RC, Eke PI. Case Definitions for Use in Population-Based Surveillance of Periodontitis. J Periodontol. 2007 Jul;78 Suppl 7S:1387-1399. doi: 10.1902/jop.2007.060264. PMID 29539084
- [Background] Seymour GJ, Taylor JJ. Shouts and whispers: An introduction to immunoregulation in periodontal disease. Periodontol 2000. 2004;35:9-13. doi: 10.1111/j.0906-6713.2004.003555.x. No abstract available. PMID 15107054
- [Background] Mattila VM, Raisamo S, Pihlajamaki H, Mantysaari M, Rimpela A. Sports activity and the use of cigarettes and snus among young males in Finland in 1999-2010. BMC Public Health. 2012 Mar 22;12:230. doi: 10.1186/1471-2458-12-230. PMID 22439614
- [Background] Mundel T. Nicotine: Sporting Friend or Foe? A Review of Athlete Use, Performance Consequences and Other Considerations. Sports Med. 2017 Dec;47(12):2497-2506. doi: 10.1007/s40279-017-0764-5. PMID 28791650
- [Background] Siddiqi K, Shah S, Abbas SM, Vidyasagaran A, Jawad M, Dogar O, Sheikh A. Global burden of disease due to smokeless tobacco consumption in adults: analysis of data from 113 countries. BMC Med. 2015 Aug 17;13:194. doi: 10.1186/s12916-015-0424-2. PMID 26278072
- [Background] Carlsson S, Andersson T, Araghi M, Galanti R, Lager A, Lundberg M, Nilsson P, Norberg M, Pedersen NL, Trolle-Lagerros Y, Magnusson C. Smokeless tobacco (snus) is associated with an increased risk of type 2 diabetes: results from five pooled cohorts. J Intern Med. 2017 Apr;281(4):398-406. doi: 10.1111/joim.12592. Epub 2017 Feb 6. PMID 28164394
- [Background] Genco RJ, Borgnakke WS. Risk factors for periodontal disease. Periodontol 2000. 2013 Jun;62(1):59-94. doi: 10.1111/j.1600-0757.2012.00457.x. PMID 23574464
- [Background] Heikkinen AM, Pajukanta R, Pitkaniemi J, Broms U, Sorsa T, Koskenvuo M, Meurman JH. The effect of smoking on periodontal health of 15- to 16-year-old adolescents. J Periodontol. 2008 Nov;79(11):2042-7. doi: 10.1902/jop.2008.080205. PMID 18980511
- [Background] Natvig Norderhaug I, Dybing E, Gilljam H, Lind PO, Lund KE, Morland J, Stegmayr B, Hofmann B, Orjasaeter Elvsaas IK. Health Effects and Dependency Associated with Snuff Consumption [Internet]. Oslo, Norway: Knowledge Centre for the Health Services at The Norwegian Institute of Public Health (NIPH); 2005 Jun. Report from Norwegian Knowledge Centre for the Health Services (NOKC) No. 06-2005. Available from http://www.ncbi.nlm.nih.gov/books/NBK464770/ PMID 29319988
- [Background] Hugoson A, Rolandsson M. Periodontal disease in relation to smoking and the use of Swedish snus: epidemiological studies covering 20 years (1983-2003). J Clin Periodontol. 2011 Sep;38(9):809-16. doi: 10.1111/j.1600-051X.2011.01749.x. Epub 2011 Jul 18. PMID 21762421
- [Background] Bergstrom J, Keilani H, Lundholm C, Radestad U. Smokeless tobacco (snuff) use and periodontal bone loss. J Clin Periodontol. 2006 Aug;33(8):549-54. doi: 10.1111/j.1600-051X.2006.00945.x. PMID 16899097
- [Background] Lee PN. Epidemiological evidence relating snus to health--an updated review based on recent publications. Harm Reduct J. 2013 Dec 6;10:36. doi: 10.1186/1477-7517-10-36. PMID 24314326
- [Background] Timberlake DS, Nikitin D, Johnson NJ, Altekruse SF. A longitudinal study of smokeless tobacco use and mortality in the United States. Int J Cancer. 2017 Jul 15;141(2):264-270. doi: 10.1002/ijc.30736. Epub 2017 Apr 24. PMID 28411395
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] GREENE JC, VERMILLION JR. THE SIMPLIFIED ORAL HYGIENE INDEX. J Am Dent Assoc. 1964 Jan;68:7-13. doi: 10.14219/jada.archive.1964.0034. No abstract available. PMID 14076341
- [Background] Soder PO, Jin LJ, Soder B, Wikner S. Periodontal status in an urban adult population in Sweden. Community Dent Oral Epidemiol. 1994 Apr;22(2):106-11. doi: 10.1111/j.1600-0528.1994.tb01582.x. PMID 8205774
- [Background] Soder B, Jin LJ, Soder PO, Wikner S. Clinical characteristics of destructive periodontitis in a risk group of Swedish urban adults. Swed Dent J. 1995;19(1-2):9-15. PMID 7597634
- [Background] Henley SJ, Thun MJ, Connell C, Calle EE. Two large prospective studies of mortality among men who use snuff or chewing tobacco (United States). Cancer Causes Control. 2005 May;16(4):347-58. doi: 10.1007/s10552-004-5519-6. PMID 15953977
- [Background] An N, Andrukhov O, Tang Y, Falkensammer F, Bantleon HP, Ouyang X, Rausch-Fan X. Effect of nicotine and porphyromonas gingivalis lipopolysaccharide on endothelial cells in vitro. PLoS One. 2014 May 12;9(5):e96942. doi: 10.1371/journal.pone.0096942. eCollection 2014. PMID 24820118
- [Background] Benowitz NL. Nicotine and smokeless tobacco. CA Cancer J Clin. 1988 Jul-Aug;38(4):244-7. doi: 10.3322/canjclin.38.4.244. PMID 3135084
- [Background] Tanner T, Kamppi A, Pakkila J, Jarvelin MR, Patinen P, Tjaderhane L, Anttonen V. Association of smoking and snuffing with dental caries occurrence in a young male population in Finland: a cross-sectional study. Acta Odontol Scand. 2014 Nov;72(8):1017-24. doi: 10.3109/00016357.2014.942877. Epub 2014 Aug 20. PMID 25141188
- [Background] Engstrom K, Magnusson C, Galanti MR. Socio-demographic, lifestyle and health characteristics among snus users and dual tobacco users in Stockholm County, Sweden. BMC Public Health. 2010 Oct 18;10:619. doi: 10.1186/1471-2458-10-619. PMID 20955584
- [Background] Norberg M, Malmberg G, Ng N, Brostrom G. Who is using snus? - Time trends, socioeconomic and geographic characteristics of snus users in the ageing Swedish population. BMC Public Health. 2011 Dec 14;11:929. doi: 10.1186/1471-2458-11-929. PMID 22169061